CLINICAL TRIAL: NCT00297427
Title: Efficacy of Acupuncture in Treating Urinary Incontinence
Brief Title: Acupuncture for Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sandra Engberg, Professor and Associate Dean for Graduate Clinical Education, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AT002175-01A1 (NIH); R01AT002175-01A1 (NIH); NCT00177450 (obsolete NCT alias)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Subjects will 12 acupuncture treatments over 6 weeks; treatment sessions occur twice a week. A total of 12 acupuncture needles will be inserted bilaterally at two leg points and four back points. Needles are manually inserted through a standard guide tube contained within a fitted sheath and the basal ring secured to the skin by double-sided tape. The needles remain in place for 25 minutes and are manually stimulated twice during each treatment.
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): Subjects will receive 12 sham acupuncture treatments (delivered twice a week) over 6 weeks. The sham needle is blunted needle whose shaft telescopes into the handle when tapped. While the needle appears to have been inserted, it does not actually penetrate the skin. It is held in place by the same standard guide tube used in the true acupuncture group. The acupuncture points and duration of treatment are the same as for the true acupuncture group.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture twice weekly for 6 weeks.
  Arms: Acupuncture
Other: Sham acupuncture — Twice a week for 6 weeks
  Arms: Sham acupuncture

SUMMARY:
This research study will evaluate the effectiveness of acupuncture in decreasing urinary incontinence (involuntary urine loss) in women. The study will involve 12 acupuncture sessions over 6 weeks. We will compare the effectiveness of acupuncture and sham (placebo) acupuncture (a procedure in which the needle feels like it penetrates the skin, but is not actually inserted into the body) on the frequency and volume of involuntary (accidental) urine loss after completing the intervention, and again one month later. Individuals participating in this study will be randomly assigned to receive either the actual or sham acupuncture. Randomization means being assigned by chance, similar to flipping a coin. Study participants will not know which group (actual or sham acupuncture) they were assigned to until one month after completing the 6-weeks of treatment. The sham acupuncture needles look similar to the real acupuncture needles and feel like they penetrate the skin, but do not actually do so. If individuals are assigned to the sham acupuncture group, they will be eligible to receive the actual acupuncture one month after completing the sham acupuncture if they wanted to. All individuals will be followed for 6 months after completing the acupuncture treatments.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Urge or stress urinary incontinence at least twice a week on average for at least 3 months

Exclusion Criteria:

* History of previous acupuncture
* History of a neurologic problem such as Parkinson's disease or multiple sclerosis that could affect bladder function
* Current treatment with overactive bladder medications or medications that relax the bladder
* Urinary catheter
* Pregnancy
* Inability to empty the bladder effectively
* Inability to toilet independently
* Current treatment with steroid
* Interstitial cystitis
* Chronic pelvic pain
* Current treatment with warfarin

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Engberg, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: Initial Intervention
Arm/Group | Acupuncture | Sham Acupuncture
Started | 64 (Intention-to-treat analysis; all randomized subjects were included in analysis) | 63 (Intention-to-treat analysis; all randomized subjects were included in analysis)
Completed | 56 | 54
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Death | 0 | 1
Period: Phase 2: Optional Crossover for Sham
Arm/Group | Acupuncture | Sham Acupuncture
Started | 54 | 0 (There was no cross-over to sham acupuncture as this was a wait list control design)
Crossed Over to True Acupuncture | 42 (54 subjects completed the sham acupuncture & were offered the opportunity to cross-over; 12 declined) | 0 (There was no cross-over to sham acupuncture as this was a wait list control design)
Completed | 38 | 0 (There was no cross-over to sham acupuncture as this was a wait list control design)
Not Completed | 16 | 0
Not completed — Withdrawal by Subject | 15 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Phase 3: Follow-up Post-True Acupuncture
Arm/Group | Acupuncture | Sham Acupuncture
Started | 94 | 0 (Only subjects who received true acupuncture initially or after cross-over entered follow-up)
Completed | 60 (Subjects who completed=/>1 follow-up visits and were evaluated for booster acupuncture) | 0 (Only subjects who received true acupuncture initially or after cross-over entered follow-up)
Not Completed | 34 | 0
Not completed — Withdrawal by Subject | 29 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Could not complete outcome diary | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.31 (11.93) | 57.41 (11.86) | 56.86 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 63 | 125
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 50 | 57 | 107
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 0 | 2
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 29.47 (6.68) | 29.54 (6.65) | 29.50 (6.64)
Co-morbidities [Mean (Standard Deviation); unit: co-morbid health problems] — Number of co-morbid health problems
  co-morbid health problems | 2.92 (2.37) | 2.82 (2.09) | 2.87 (2.23)
Number of prescription medications [Mean (Standard Deviation); unit: Prescription medications] — Number of prescription medications taken on a regular basis
  Prescription medications | 2.20 (2.2) | 2.22 (2.33) | 2.21 (2.26)
Vaginal deliveries [Mean (Standard Deviation); unit: Vaginal deliveries] — Number of vaginal deliveries
  Vaginal deliveries | 1.59 (1.51) | 1.43 (1.24) | 1.51 (1.38)
Menopausal Status [Number; unit: participants] — Number of women in each group who self-reported cessation of menses
  participants
    Postmenopausal | 41 | 43 | 84
    Premenopausal | 23 | 20 | 43
Hormone replacement therapy [Number; unit: participants] — Number of women taking hormone replacement therapy
  participants
    Yes | 7 | 7 | 14
    No | 34 | 36 | 70
    No applicable (premenopausal) | 23 | 20 | 43
Limited mobility [Number; unit: participants] — Number of women with self-reported limitations in mobility
  participants
    Yes | 8 | 9 | 17
    No | 56 | 54 | 110
Incontinent episodes/day [Mean (Standard Deviation); unit: episodes/day] — Episodes of urinary incontinence per day as measured by bladder diary
  episodes/day | 2.19 (1.57) | 2.59 (2.12) | 2.39 (1.87)
Duration of urinary incontinence [Mean (Standard Deviation); unit: Years] | 9.81 (9.08) | 8.61 (9.98) | 9.22 (9.52)
Mental Health-Related Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Medical Outcomes Short Form-36 (SF-36) where higher scores indicate better quality of life. The possible score range is 0 to 100.
  units on a scale | 55.49 [48.03 to 58.99] | 55.90 [49.22 to 60.52] | 55.67 [49.22 to 59.42]
Physical Health-Related Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Medical Outcomes Study Short Form-36 (SF-36) where higher scores indicate better quality of life. Possible score range is 0 to 100.
  units on a scale | 54.32 [48.03 to 57.19] | 53.83 [48.47 to 56.80] | 54.17 [48.34 to 57.08]
Incontinence-Specific Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Incontinence Impact Questionnaire total score. Possible scores range from 0 to 300 with higher scored indicating worse urinary-specific quality of life.
  units on a scale | 55.95 [27.94 to 121.88] | 61.43 [20.63 to 118.78] | 57.78 [25.56 to 118.78]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Incontinent Episodes
Description: Percent change in incontinent episodes (measured by self-report electronic bladder diary) at 1 week post-intervention (true or sham acupuncture) relative to baseline.
Time Frame: Baseline to 1 Week post-intervention
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: percent change in incontinent episodes
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percent change in incontinent episodes | -38.26 (42.63) | -15.29 (65.41)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Primary Outcome: Percent Change in Incontinent Episodes
Description: Percent change in incontinent episodes (measured by self-report electronic bladder diary) 4 weeks post true or sham acupuncture
Time Frame: 4 weeks post true or sham acupuncture
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: percent change in incontinent episodes
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percent change in incontinent episodes | -42.49 (40.24) | -34.47 (49.98)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.32, t-test, 2 sided

3. Primary Outcome: Physical Health-Related Quality of Live
Description: Percent change in physical health related quality of life measured at 1 week post-intervention (true or sham acupuncture) relative to baseline; measured by the Medical Outcomes Study Short Form-36 (SF-36) Physical Component score. Higher SF-36 Physical Component scores are considered a better outcome.
Time Frame: 1 Week post-intervention
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: percentage change relative to baseline
Groups:
- Acupuncture: True acupuncture twice a week for 6 weeks
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 0 [-3.78 to 7.29] | 0 [-6.70 to 3.35]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Physical Health-Related Quality of Life
Description: Percent change in physical health related quality of life measured at 4 weeks post intervention (true or sham acupuncture) relative to baseline; measured by the Medical Outcomes Study Short Form-36 (SF-36) Physical Component score. Positive change indicates an increase in physical health-related quality of life.
Time Frame: 4-weeks post-intervention
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: percentage change relative to baseline
Groups:
- Acupuncture: Ture acupuncture twice a week for 6 weeks
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 0.37 [-2.12 to 10.73] | 0 [-4.42 to 4.43]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Mental Health Related Quality of Life
Description: Percent change in mental health related quality of life measured at 1 week1 post intervention (true or sham acupuncture) relative to baseline; measured by the Medical Outcomes Study Short Form-36 (SF-36) Mental Health Component score. Higher Mental Health Component scores are considered a better outcome.
Time Frame: 1 week post-intervention
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: percentage change relative to baseline
Groups:
- True Acupuncture: True Acupuncture twice weekly for 6 weeks.
- Sham Acupuncture: Sham acupuncture twice weekly for 6 weeks
Arm/Group | True Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 0 [-5.71 to 7.29] | 2.66 [0 to 8.76]

6. Primary Outcome: Mental Health Related Quality of Life
Description: Percent change in mental health related quality of life measured at 4 weeks post intervention (true or sham acupuncture) relative to baseline; measured by the Medical Outcomes Study Short Form-36 (SF-36) Mental Health Component score.
Time Frame: 4 weeks post true or sham acupuncture
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: percentage change relative to baseline
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 0 [-5.59 to 3.58] | 1.81 [-0.18 to 5.17]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Incontinence-Specific Quality of Life
Description: Percent change in incontinence specific quality of life at 1 week post intervention (true or sham acupuncture) as measured by the Incontinence Impact Questionnaire. Positive values indicate improvement in incontinence-specific quality of life.
Time Frame: 1 Week post-intervention
Population: Intention-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: percentage change relative to baseline
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 26.02 [0.84 to 69.03] | 17.36 [0.53 to 48.61]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Incontinence-Specific Quality of Life
Description: Percent change in incontinence-specific quality of life a 4 weeks post-intervention (true or sham acupuncture) measured by the Incontinence Impact Questionnaire. Positive changes indicate improvement in incontinence-specific quality of life.
Time Frame: 4-weeks post-intervention
Population: Intention-to-treat
Measure: Mean (Inter-Quartile Range); unit: percentage change relative to baseline
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 64 | 63
percentage change relative to baseline | 48.01 [-6.49 to 83.40] | 32.04 [-16.84 to 65.49]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Duration of Any Beneficial Effects
Description: Time to relapse in months of participants who completed true acupuncture initially or who crossed-over following sham (offered to all sham participants)
Time Frame: monthly during follow-up up to 6 months
Population: Subjects who received true acupuncture and completed at least a 1-month follow-visit post acupuncture
Measure: Mean (Standard Error); unit: Months
Arm/Group | Acupuncture
Number analyzed (Participants) | 60
Months | 2.17 (0.25)

10. Secondary Outcome: Change in Bladder Capacity
Description: Measured by filling the bladder with sterile fluid until until the subject reported a strong urge to urinate.
Time Frame: Change from baseline to 4 weeks post-intervention
Population: Subjects who agreed to have a cystometrogram at baseline and 4 weeks after completing acupuncture or sham acupuncture.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 23 | 19
milliliters | 60.45 (114.91) | -17.89 (121.68)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.04, Repeated measures using GEE

11. Secondary Outcome: Urodynamic Diagnostic Impression of Stress Urinary Incontinence
Description: Documentation of a diagnostic impression of stress urinary incontinence following urodynamics
Time Frame: Baseline and 4 weeks post-treatment
Measure: Number; unit: participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 23 | 19
participants
  Baseline | 16 | 6
  4 weeks post-intervention | 4 | 5
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.01, Repeated measures using GEE

12. Secondary Outcome: Urodynamic Impression of Urge Urinary Incontinence
Description: Documentation of a diagnostic impression of urge urinary incontinence following urodynamics
Time Frame: Baseline and 4 weeks post true or sham acupuncture
Measure: Number; unit: participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 23 | 19
participants
  Baseline | 13 | 13
  4-weeks post intervention | 13 | 10
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.41, Repeated measures using GEE

13. Secondary Outcome: Characteristics of Responders Based on Glasses/Cups Per Day of Non-caffeinated Fluids (Including Water)
Description: Glasses/cups per day of non-caffeinated fluids (including water) at baseline
Time Frame: Baseline
Population: Responders were subjects who achieved a 50% reduction in urinary incontinent episodes by 4 weeks post true acupuncture (as their initial or relayed intervention)
Measure: Mean (Standard Deviation); unit: Glasses/cups per day
Groups:
- Responders: 50% or greater reduction in incontinent episodes following true acupuncture
- Non-responders: Less than a 50% reduction in incontinent episodes following true acupuncture
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 42 | 58
Glasses/cups per day | 6.88 (3.054) | 5.45 (2.663)
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 0.04, t-test, 2 sided — Bivariate (unadjusted) analysis
Statistical Analysis 2: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.208, 95% CI 2-sided [1.039 to 1.405] — These are the adjusted results of a multivariate logistic regression

14. Secondary Outcome: Characteristics of Responders: Duration of Urinary Incontinence (UI) in Years
Description: Duration of urinary incontinence in years
Time Frame: Baseline
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 42 | 58
years | 6.93 (6.69) | 10.66 (9.42)
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 0.023, t-test, 2 sided — This is the result from the bivariate (unadjusted) analysis
Statistical Analysis 2: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 0.030, Regression, Logistic; Odds Ratio (OR) = 0.936, 95% CI 2-sided [0.881 to 0.994] — These are the adjusted results from a multivariate logistic regression analysis

15. Secondary Outcome: Adherence to Treatment Protocol
Description: Percentage of acupuncture (true or sham) visits completed as scheduled
Time Frame: 6 weeks
Population: True and sham acupuncture subjects who completed the 6 weeks of treatment; participants who dropped out of the study during treatment were not included in this analysis
Measure: Mean (Standard Deviation); unit: percent of visits
Groups:
- Acupuncture: Acupuncture: True acupuncture twice weekly for 6 weeks
- Sham Acupuncture: Sham acupuncture twice a week for 6 weeks
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 56 | 54
percent of visits | 91.88 (9.39) | 91.05 (9.28)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

16. Secondary Outcome: Burden Associated With the Acupuncture Treatment Protocol
Description: Subjects' report of burden (difficulty) associated with the frequency, number and duration of treatment) and the position they had to remain in during the true and sham treatments. Subjects rate the difficulty associated with each of the four aspects of treatment on a 10-point scale ranging from 1 (not at all difficult) to 10 (extremely difficult). The burden score was calculated as the average of the scores on the 4 items with a possible range of 1 to 10 with higher scores indicating greater burden.
Time Frame: 1 week post-treatment
Population: The number of participants analyzed for this outcome was only those who completed the treatment protocol and the 1-week post-treatment visit. For this reason, the number is smaller than the number for the primary outcomes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 53 | 52
units on a scale | 2.25 [1.50 to 3.25] | 2.25 [1.56 to 3.50]
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Need for Booster Acupuncture During Follow-up
Description: The number of participants who were received true acupuncture (as their initial intervention or after initially receiving sham acupuncture) and were eligible to receive a booster (had a 50% or greater reduction in incontinent episodes following true acupuncture) and completed at least one month of follow-up and experienced a 30% or greater increase in incontinent episodes during follow up.
Time Frame: Monthly during the 6 month follow-up period
Population: Participants who completed true acupuncture (as either their initial treatment or following sham acupuncture), had a 50% or greater reduction in incontinent episodes at 1 or 4 weeks post-true acupuncture, and completed at least one month of follow-up.
Measure: Number; unit: participants
Arm/Group | Acupuncture
Number analyzed (Participants) | 51
participants | 43

18. Secondary Outcome: Response to Booster Acupuncture if Needed
Description: Change in the number of incontinent episodes per day following booster acupuncture
Time Frame: After the booster sessions
Population: Participants who received booster acupuncture treatments during follow-up
Measure: Mean (Standard Deviation); unit: incontinent episodes/day
Arm/Group | Acupuncture
Number analyzed (Participants) | 35
incontinent episodes/day
  Prior to booster acupuncture | 1.37 (0.97)
  Following booster acupuncture | 0.77 (0.69)
Statistical Analysis 1: Comparison: Acupuncture; Test type: Superiority or Other; p < .001, t-test, 1 sided

19. Secondary Outcome: Pelvic Floor Muscle Strength
Description: Change in average duration of pelvic floor muscle contraction measured by electromyography. Subjects were instructed to tighten their pelvic floor muscles when prompted and hold the contraction until told to relax (up to 10 seconds). This was repeated three times and the duration of the contraction time was averaged.
Time Frame: Baseline and 1 week post true or sham acupuncture
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 45 | 45
seconds | 0.78 (4.66) | 0.04 (5.02)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.48, t-test, 2 sided

20. Secondary Outcome: Pelvic Floor Muscle Strength
Description: as for outcome 19
Time Frame: Baseline and 4 weeks post true or sham acupuncture
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 41 | 42
seconds | 0.71 (4.98) | 0.53 (4.01)
Statistical Analysis 1: Comparison: Acupuncture vs Sham Acupuncture; Test type: Superiority or Other; p = 0.86, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6-weeks; during the intervention period (true and sham acupuncture) adverse events were assessed after each intervention visit
Description: After each visit subjects completed an investigator-developed acupuncture symptom questionnaire. Questions were based on a review of literature reporting adverse effects during acupuncture. Subjects were included if they completed at least one adverse event questionnaire.
Arm/Group | Acupuncture | Sham Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 56/63 | 48/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=63) | Sham Acupuncture (N=63)
Fatigue (General disorders) | 21 | 16 — Reported feeling tired during or after at least one acupuncture (true or sham) treatment
Drowsy (General disorders) | 17 | 15 — Reported feeling drowsy during or after at least acupuncture (true or sham) treatment
Increase in incontinent episodes (Renal and urinary disorders) | 26 | 21 — Reported experiencing an increase in urinary incontinent episodes after at least one acupuncture (true or sham) treatment
Increase in urinary urgency (Renal and urinary disorders) | 20 | 18 — Reported an increase in urinary urgency after at least one acupuncture (true or sham) treatment
Increase in stress urinary incontinence (Renal and urinary disorders) | 23 | 15 — Reported an increase in urinary leakage with physical activity after at least one acupuncture (true or sham) treatment
Itching at acupuncture site (Skin and subcutaneous tissue disorders) | 21 | 16 — Reported itching at the acupuncture site after at least one acupuncture (true or sham) treatment
Dizzy (General disorders) | 8 | 9 — Reported feeling dizzy during or after at least one acupuncture (true or sham) treatment
Bleeding at acupuncture site (Blood and lymphatic system disorders) | 41 | 2 — Reported any bleeding at any of the acupuncture sites during or after an acupuncture (true or sham) treatment
Pain during treatment (General disorders) | 51 | 22 — Pain during needle insertion reported during at least one acupuncture (true or sham) treatment
Aching at needle insertion site(s) (General disorders) | 41 | 14 — Reported aching at any needle insertion site after at least one acupuncture (true or sham) treatment
Bruising (Blood and lymphatic system disorders) | 27 | 4 — Reported bruising at a needle insertion site after at least one acupuncture (true or sham) treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No